CLINICAL TRIAL: NCT02448147
Title: Interval Training Versus Continuous Training on Peripheral Perfusion and Sympathetic Activity in Patients With Heart Failure
Brief Title: Interval Versus Continuous Training in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Guilherme Veiga Guimarães,, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/08990-1
Record Dates: First submitted 2015-05-11; First posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Heart Failure
Keywords: Heart failure; Exercise; Biomarkers; Sympathetic Nervous System; MicroRNA
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interval training (Active Comparator)
  Interventions: Behavioral: Interval training
- Continuous training (Active Comparator)
  Interventions: Behavioral: Continuous training
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Interval training — Patients will be submitted to three months aerobic exercise training, three times per week. Each session will have two levels of intensity: one minute at respiratory compensation point heart rate intercalating with two minutes at anaerobic threshold heart rate during thirty minutes.
  Other Names: Interval exercise training; Interval exercise
  Arms: Interval training
Behavioral: Continuous training — Patients will be submitted to three months aerobic exercise training, three times per week. Each session will have only one level of intensity during stimulus phase of exercise, lasting thirty minutes: heart rate (HR) target is defined as 1/3x(HR at respiratory compensation point) + 2/3x(HR anaerobic threshold)
  Other Names: Continuous exercise training; Continuous exercise
  Arms: Continuous training

SUMMARY:
BACKGROUND: The physiopathology of the heart failure involves compensatory mechanisms as exacerbated neurohormonal activity, endothelial dysfunction and consequently the muscle disability and exercise intolerance. The interval exercise training has been proposed as one efficient method to heart failure patients. It seems that the main mechanism involved in the benefit of the interval exercise training is "shear stress". AIM: To study the interval exercise training versus the continuous exercise training in the sympathetic activity and in the peripheral muscle perfusion in heart failure patients. Moreover, we will evaluate the muscle apoptosis, microRNA in plasma and muscle biopsy, biomarkers levels of inflammation, quality of life and exercise capacity. METODOLOGY: Will be selected 40 patients (male and female) with age between 30 and 60 years, left ventricular ejection fraction less than 40% and functional class I, II and III. These patients will be randomized into three groups: Interval (AIT), continuous (MCT) and control (CG). All patients will be evaluated with microneurography, peripheral muscle perfusion, muscle biopsy, blood samples, accelerometer, cardiopulmonary exercise test and quality of life before and after end of the period of 03 (three) months.

ELIGIBILITY:
Inclusion Criteria:

* stable chronic heart failure without changing in treatment for at least 6 weeks
* ejection fraction less then 40%, as measured by transthoracic echocardiography
* optimal clinical treatment for chronic heart failure according to current guidelines.

Exclusion Criteria:

* asthma or chronic obstructive pulmonary disease using inhaled corticosteroids
* functional class IV (New York Heart Association - NYHA)
* atrial fibrillation
* complex ventricular arrhythmia
* pacemaker or implantable cardioversor/defibrillators
* chronic renal insufficiency, defined as serum creatinine above 2,5 mg/dL
* intermittent claudication
* morbid obesity
* cirrhosis
* alcoholism
* using illicit drugs
* performing regular physical activity
* participating in another study
* invasive procedure planned
* persistent nonadherence to therapeutic regimen
* peak respiratory exchange ratio (RER) lower than 1.00

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Muscular sympathetic nervous activity | 12 weeks
  Muscular sympathetic nervous activity was measured by in peroneal nerve microneurography.
Peripheral muscular perfusion | 12 weeks
  Peripheral muscular perfusion was measured by near-infrared spectroscopy (NIRS) above vastus lateral muscle during exercise.
Biomarkers | 12 weeks
  Serum levels of biomarkers of inflammation (interleukin-6, tumor necrosis factor alpha and adiponectin) and fibrosis (galectin-3).

SECONDARY OUTCOMES:
Daily life physical activity | 12 weeks
  Daily life physical activity determined by Baecke physical activity questionnaire and by a triaxial digital accelerometer during 24 hs.
MicroRNA | 12 weeks
  Blood levels of selected microRNAs

CONTACTS AND LOCATIONS:
Overall Officials: Miguel MF Silva, MD, Study Chair — Heart Institute (InCor) HC FMUSP; Guilherme V Guimaraes, PhD, Principal Investigator — Heart Institute (InCor) HC FMUSP
Locations (1):
- Heart Institute - São Paulo University School of Medicine, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Fernandes-Silva MM, Guimaraes GV, Rigaud VO, Lofrano-Alves MS, Castro RE, de Barros Cruz LG, Bocchi EA, Bacal F. Inflammatory biomarkers and effect of exercise on functional capacity in patients with heart failure: Insights from a randomized clinical trial. Eur J Prev Cardiol. 2017 May;24(8):808-817. doi: 10.1177/2047487317690458. Epub 2017 Jan 30. PMID 28134562